CLINICAL TRIAL: NCT01009372
Title: Prospective Study on the Effects of the Intermittent Pneumoperitoneum (IPP) Work Break Scheme on Surgeons and Patients.
Brief Title: The Intermittent Pneumoperitoneum Scheme of Work Breaks in Complex Laparoscopic Surgery
Acronym: IPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Technische Universität Dresden (Other); University of Zurich (Other)
Responsible Party: Carsten Engelmann, Consultant Surgeon, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IPP 67; 4165; 3-2-2006 (Other: Ethical Commission Hannover Medical School, 30625 Hannover)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: Stress Physiology; Staff Work Load; Artificial Pneumoperitoneum; Anuria
Keywords: surgeon's physiology; stress response; break scheme
MeSH Terms: conditions — Anuria; Fractures, Stress | interventions — indolepropanol phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- breaks during laparoscopic surgery (Experimental): Intraoperative Breaks were instituted in the intervention group. The other group operated conventionally without breaks
  Interventions: Behavioral: IPP

INTERVENTIONS:
Behavioral: IPP — Institution of intraoperative breaks for the surgeon with release of pneumoperitoneum for patient
  Other Names: break schemes

SUMMARY:
Many people spanning from air traffic controllers to simple production line workers share regular compulsive breaks to revert fatigue whilst they work. This is uncommon for medical operators - a macho image is still as prevalent in real life as it is in countless TV series.

We report on the first clinical trial on regular intraoperative breaks. For one time we turned our scientific curiosity to ourselves. This included the intraoperative collection of body fluids and required transparency which was not easy to obtain. It was rewarded with striking results: Regular intraoperative breaks lowered significantly the operators stress hormone levels, improved error-performance testing results and musculoskeletal fatigue scores. Subjectively the breaks enhanced the practitioners satisfaction.

Surprisingly the operator's breaks were not at the cost of the patient: because the did not prolong the overall operation time at all and - in our setting- they significantly increased of cardiac output and urine production.

DETAILED DESCRIPTION:
Abstract

Background: Work breaks at close intervals are common in fields with high workload but not yet for medical operators. We evaluated the effects of intraoperative breaks (five minutes every half hour) on the surgeon and on the patient.

Methods: Operations were randomized to either a scheme with intraoperative breaks and release of the pneumoperitoneum (intermittent pneumoperitoneum = IPP) or a conventional conduct (CPP). Stress hormones and α-amylase were determined in the surgeon's saliva pre-, intra- and postoperatively. Mental performance and error scores, musculoskeletal strain and continuous ECG were secondary endpoints. The children's physiology was monitored.

Findings:

Regular intraoperative breaks did not prolong the operation. The surgeon's cortisol levels during the operation were reduced. There were fewer intraoperative events in the IPP vs. the CPP group. The pre- to postoperative increase in the error rates of the bp-concentration test was reduced in the IPP group. The relevant locomotive strain-scores were reduced by IPP.

There was no negative impact on the patient. Interpretation: Our data support the idea that work breaks during complex laparoscopic surgery can reduce psychological stress and preserve performance with at least similar patient outcome compared to the traditional work scheme.

ELIGIBILITY:
Inclusion Criteria:

* complex laparoscopic operations in children (duration > 100 minutes)

Exclusion Criteria:

* age under 4 weeks
* operations which had to be performed in an open surgery mode

Ages: 4 Weeks to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
hormonal stress response of the operating surgeon: cortisol, amylase, testosterone, dehydroepiandrosterone (DHEA) | 1 day

SECONDARY OUTCOMES:
continuous ECG, concentration and performance (bp-test ), Self ratings of own satisfaction, performance, musculoskeletal system (MSS) and ophthalmologic strain | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Benno M Ure, PhD, Study Director — Hannover Medical School, 30625 Hannover
Locations (1):
- Hannover Medical School, Pediatric Surgery, Hanover, Lower Saxony, Germany

REFERENCES:
- [Background] Kumari M, Badrick E, Chandola T, Adam EK, Stafford M, Marmot MG, Kirschbaum C, Kivimaki M. Cortisol secretion and fatigue: associations in a community based cohort. Psychoneuroendocrinology. 2009 Nov;34(10):1476-85. doi: 10.1016/j.psyneuen.2009.05.001. Epub 2009 Jun 3. PMID 19497676